CLINICAL TRIAL: NCT04421222
Title: A Phase 1, Open-label Study to Evaluate the Safety, Pharmacokinetics, and Anti-Tumor Activity of Oral EPI-7386 in Patients with Castration-Resistant Prostate Cancer
Brief Title: Oral EPI-7386 in Patients with Castration-Resistant Prostate Cancer
Acronym: EPI-7386
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated early due to a lack of improved efficacy.
Sponsor: ESSA Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPI-7386-CS-001
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BID protein, human; Abiraterone Acetate; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Part A/Phase 1a: Cohort 1 (Completed) (Experimental): 200 mg EPI-7386
  Interventions: Drug: EPI-7386 (QD)
- Part A/Phase 1a: Cohort 2 (Completed) (Experimental): 400 mg EPI-7386
  Interventions: Drug: EPI-7386 (QD)
- Part A/Phase 1a: Cohort 3 (Completed) (Experimental): 600 mg EPI-7386
  Interventions: Drug: EPI-7386 (QD)
- Part A/Phase 1a: Cohort 4 (Completed) (Experimental): 800 mg EPI-7386
  Interventions: Drug: EPI-7386 (QD)
- Part A/Phase 1a: Cohort 5 (Completed) (Experimental): 1000 mg EPI-7386
  Interventions: Drug: EPI-7386 (QD)
- Part A/Phase 1a: Cohort 6 (Completed) (Experimental): 800 mg EPI-7386
  Interventions: Drug: EPI-7386 (BID)
- Part A/Phase 1a: Cohort 7 (Completed) (Experimental): 1200 mg EPI-7386
  Interventions: Drug: EPI-7386 (BID)
- Part A/Phase 1b: Cohort 1 (Completed) (Experimental): 600 mg EPI-7386 BID
  Interventions: Drug: EPI-7386 (BID)
- Part A/Phase 1b: Cohort 2 (Experimental): 600 mg EPI-7386 QD
  Interventions: Drug: EPI-7386 (QD)
- Part B/Cohort 1a (Experimental): 600 mg EPI-7386 + 1000 mg Abiraterone Acetate + Prednisone
  Interventions: Drug: EPI-7386 (QD); Drug: Abiraterone acetate
- Part B/Cohort 1b (Experimental): 800 mg EPI-7386 + 1000 mg Abiraterone Acetate + Prednisone
  Interventions: Drug: EPI-7386 (QD); Drug: Abiraterone acetate
- Part B/Cohort 1c (Experimental): 1200 mg EPI-7386 + 1000 mg Abiraterone Acetate + Prednisone
  Interventions: Drug: EPI-7386 (BID); Drug: Abiraterone acetate
- Part B/Cohort 2a (Experimental): 600 mg EPI-7386 monotherapy for 12 weeks then 600 mg EPI-7386 + 240 mg Apalutamide
  Interventions: Drug: EPI-7386 (QD); Drug: Apalutamide
- Part B/Cohort 2b (Experimental): 800 mg EPI-7386 monotherapy for 12 weeks then 800 mg EPI-7386 + 240 mg Apalutamide
  Interventions: Drug: EPI-7386 (QD); Drug: Apalutamide
- Part B/Cohort 2c (Experimental): 1200 mg EPI-7386 monotherapy for 12 weeks then 1200 mg EPI-7386 + 240 mg Apalutamide
  Interventions: Drug: EPI-7386 (BID); Drug: Apalutamide

INTERVENTIONS:
Drug: EPI-7386 (QD) — Once daily oral dose of EPI-7386
  Arms: Part A/Phase 1a: Cohort 1 (Completed); Part A/Phase 1a: Cohort 2 (Completed); Part A/Phase 1a: Cohort 3 (Completed); Part A/Phase 1a: Cohort 4 (Completed); Part A/Phase 1a: Cohort 5 (Completed); Part A/Phase 1b: Cohort 2; Part B/Cohort 1a; Part B/Cohort 1b; Part B/Cohort 2a; Part B/Cohort 2b
Drug: EPI-7386 (BID) — Twice daily oral dose of EPI-7386
  Arms: Part A/Phase 1a: Cohort 6 (Completed); Part A/Phase 1a: Cohort 7 (Completed); Part A/Phase 1b: Cohort 1 (Completed); Part B/Cohort 1c; Part B/Cohort 2c
Drug: Abiraterone acetate — Once daily dose of abiraterone acetate
  Arms: Part B/Cohort 1a; Part B/Cohort 1b; Part B/Cohort 1c
Drug: Apalutamide — Once daily dose of apalutamide
  Arms: Part B/Cohort 2a; Part B/Cohort 2b; Part B/Cohort 2c

SUMMARY:
This is a phase I, clinical research study of EPI-7386, an investigational drug being studied as a treatment for patients with prostate cancer. All patients in the study will receive EPI-7386.

Since this is the first study of EPI-7386 in humans, there is no information about how it affects people or what dose should be used. Therefore, the main purpose of this study is to assess the safety (side effects) of EPI-7386 and to find a dose that can be given without unacceptable side effects.

There are other important things that will be evaluated during the study:

* How the amount of EPI-7386 in the blood changes over time.
* The effect of EPI-7386 on prostate cancer.
* The effect of EPI-7386 on certain substances in the body.
* The possibility that EPI-7386 can interact with other drugs.

The study will be conducted in 2 parts:

* Part A: To evaluate the safety and tolerability of EPI-7386 as a single agent via 2 Phases:

  * Phase 1a: Dose Escalation (mCRPC)
  * Phase 1b: Dose Expansion (mCRPC)
* Part B: To evaluate 2 parallel enrolling cohorts (Cohort 1 and Cohort 2) of EPI-7386 in combination of apalutamide acetate + prednisone (AAP) or apalutamide (APA):

  * Cohort 1: Combination with AAP in mHSPC or mCRPC patients
  * Cohort 2: Will evaluate the anti-tumor activity of EPI-7386 for a limited window of time (12 weeks EPI-7386 monotherapy prior to the start of combination therapy with APA) in nmCRPC patients unperturbed by previous 2nd generation anti-androgen therapies or chemotheraphy.

ELIGIBILITY:
Part A/Phase 1a (Dose Escalation) Inclusion Criteria:

* Male 18 years of age or older.
* Histologically, pathologically, or cytologically confirmed prostate cancer without small cell features.
* Evidence of castration-resistant prostate cancer (CRPC).
* Presence of metastatic disease at study entry documented by 1 or more bone lesions on bone scan or by soft tissue disease observed by CT/MRI.
* Limited further treatment options available known to confer clinical benefit in this disease setting from the perspective of the treating physician. Specifically, patients must have progressed on at least 2, but not more than 3, prior approved systemic therapies for mCRPC which include at least one, but not more than 2, second generation anti-androgen drug.
* Patients may have received prior docetaxel for mCSPC or mCRPC but must not have had disease progression during, or within 6 months of completing chemotherapy. Only one line of prior chemotherapy is allowed.
* Evidence of progressive disease defined as 1 or more Prostate Cancer Working Group 3 (PCWG3) criteria.
* The patient must have recovered from toxicities related to any prior treatments.
* Castrate at screening.
* Patients receiving bisphosphonates or other approved bone-targeting therapy must be on a stable dose for at least 4 weeks prior to the start of study drug.
* Demonstrate adequate organ function.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

Part A/Phase 1b (Dose Expansion) Inclusion Criteria:

The inclusion criteria for this cohort are the same as for Phase 1a with the exception of: limit of prior therapies to 2 and prior chemotherapy is not allowed for this cohort of patients.

Part B/Cohort 1 (EPI-7386 in combination with AAP) Inclusion Criteria:

* Patients are eligible to enroll in this cohort if they meet the clinical criteria for receiving AAP as standard of care treatment as per label (i.e., high-risk mHSPC or mCRPC).
* All other inclusion criteria listed for Part A/Phase 1a apply except for those that do not apply to mHSPC or mCRPC patients (i.e. evidence of CRPC and limited treatment options for mCRPC).

Part B/Cohort 2 (Window of Opportunity with clinical endpoints followed by combination with Apalutamide)

* Male 18 years of age or older.
* Histologically, pathologically, or cytologically confirmed prostate cancer without small cell features.
* Evidence of castration-resistant prostate cancer (CRPC).
* Patients who received a first generation anti-androgen as part of an initial combined androgen blockade therapy or as second-line hormonal therapy must show continuing disease (PSA) progression off the anti-androgen for at least 4 weeks prior to enrollment.
* At least 4 weeks must have elapsed from the use of 5-α reductase inhibitors, estrogens, and any other anti-cancer therapy prior to enrollment.
* At least 4 weeks must have elapsed from major surgery or radiation therapy prior to enrollment.
* The patient must have recovered from toxicities related to any prior treatments.
* Castrate at screening.
* Demonstrate adequate organ function.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

Part A Phase 1a and Phase 1b Exclusion Criteria:

* Biologic anti-cancer therapy or a cytotoxic chemotherapy within 4 weeks prior to the start of study drug.
* Use of hormonal agents with anti-tumor activity against prostate cancer within 4 weeks prior to the start of study drug.
* Any lutamides or abiraterone within 14 days or 5 half-lives, whichever is longer prior to start of study drug.
* Use of radium-223 dichloride or other radioligand/radiopharmaceutical within 28 days prior to the start of study drug.
* Received limited-field palliative bone radiotherapy >5 fractions and/or any radiotherapy within 2 weeks prior to the start of study drug.
* Received a blood transfusion within 28 days of screening.
* Received prior chemotherapy (for Part 1b Cohort A only).
* Known intra-cerebral disease or brain metastasis unless adequately treated and stable for the last 4 weeks before enrollment.
* Spinal cord compression.
* Diagnosis of another invasive malignancy within the previous 3 years other than curatively treated non-melanomatous skin cancer or superficial urothelial carcinoma.
* Gastrointestinal disorder affecting absorption.
* Significant cardiovascular disease.
* Concurrent disease or any clinically significant abnormality.
* Use of strong inducers of CYP3A within 14 days of the first dose of study drug.

Part A Phase 1b (Dose Expansion) Exclusion Criteria:

The exclusion criteria for this cohort are the same as the criteria from Phase 1a with the addition of the following:

• Any prior treatment with chemotherapy.

Part B Cohort 1 (EPI-7386 in combination with AAP) Exclusion Criteria:

The exclusion criteria for this cohort are the same as the criteria from Phase 1a with the addition of the following:

* Use of concomitant CYP2D6 substrates with narrow therapeutic index.
* Known allergies, hypersensitivity, or intolerance to the excipients of AA (refer to AA Investigator's Brochure [IB] or package inserts as appropriate).

Part B Cohort 2 (Window of Opportunity with clinical endpoints followed by combination with Apalutamide)

* Presence of distant metastases, including visceral, nodal and bones involvement. Exception: pelvic lymph nodes < 2 cm in short axis (N1) located below the iliac bifurcation are allowed.
* Symptomatic loco-regional disease requiring medical intervention, such as moderate or severe urinary obstruction or hydronephrosis due to primary tumor.
* Prior treatment with second generation anti-androgens.
* Prior treatment with CYP17 inhibitors.
* Prior treatment with radiopharmaceutical agents, immunotherapy, or any other investigational agent for nmCRPC.
* Prior chemotherapy.
* History or evidence of: prior malignancy (other than adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) within 3 years prior to enrollment; severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events; uncontrolled hypertension.
* Gastrointestinal disorder affecting absorption.
* Use of strong inducers of CYP3A within 14 days of the first dose of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 71 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
The primary safety variable for Part A/Phase 1a of the study is the incidence of protocol-defined DLT during the DLT assessment period (first 28 days of dosing). | 2 months
  The DLTs will be characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for AEs [NCI CTCAE version 5.0]), timing, seriousness, and relationship to study drug.
The primary efficacy variable for Part A/Phase 1b is the proportion of patients with a decline from baseline in PSA blood concentrations of ≥50% and ≥90% at any time point during daily dosing with EPI-7386. | 12 months
The primary efficacy variable for Part B/Cohort 1 is the incidence of protocol-defined DLT during the DLT assessment period (first 28 days of dosing); TEAEs; abnormalities in clinical laboratory parameters/vitals/ECGs; and changes in ECOG. | 6 months
  The DLTs will be characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for AEs [NCI CTCAE version 5.0]), timing, seriousness, and relationship to study drug.
  TEAEs and abnormalities in clinical laboratory parameters/vitals/ECGs will be characterized by type, frequency, severity, timing, seriousness and relationship to study treatment.
The primary efficacy variable for Part B/Cohort 2 is the proportion of patients with a decline from baseline in PSA blood concentrations of ≥50% and ≥90% at any time point during daily dosing with single agent EPI-7386 up to Week 12. | 4 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Comprehensive Cancer Center of NV Las Vegas, Las Vegas, Nevada
  - Great Lakes Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Canada (2):
  - BC Cancer, Vancouver, British Columbia
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No